CLINICAL TRIAL: NCT05441969
Title: In Vivo Cortical Excitability Modulation in Major Depressive Disorder
Acronym: PDM-TMS
Status: Recruiting | Type: Observational
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Principal Investigator, Albino Maia, Director of Neuropsychiatry Unit, Champalimaud Foundation, Fundacao Champalimaud
Other Study IDs: PDM-TMS
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Cortical Excitability Modulation; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Current major depressive episode group: Adult individuals (18-65 yrs) diagnosed with current major depressive episode (MDE), under treatment or medication naif, starting a new antidperessant strategy (n≈30).
  Interventions: Other: No intervention/expousure
- Maintenance antidepressant treatment group: Adult individuals (18-65 yrs) previously diagnosed with major depressive episode (MDE) currently remitted under continuation or maintenance antidepressant treatment (n≈30).
  Interventions: Other: No intervention/expousure
- Healthy subjects group: Adult individuals (18-65 yrs) without current diagnosis of major neuropsychiatric disorders, inlcluding MDE, hence not under any antidepressant medication. The same exclusion criteria will be applied as in the two clincial groups.
  Interventions: Other: No intervention/expousure

INTERVENTIONS:
Other: No intervention/expousure — No interventions/expousure since this is an observational study.

SUMMARY:
The pathophysiology of Major Depression Disorder (MDD) is unclear, with several theories for its neurobiological mechanisms. One possible explanation is the presence of altered neuroplasticity, which can be studied by Transcranial Magnetic Stimulation (TMS). Using TMS to study these mechanisms is performed by applying electromagnetic stimuli to the motor cortex, to obtain measures of temporary cortical excitability modulation. It is known that depressed patients with higher cortical modulation are more responsive to a TMS treatment course. However, it is unknown if there are differences in cortical modulation between depressed patients and healthy subjects. Our goal is to answer this question and contribute towards clarification of the neuroplasticity mechanisms underlying MDD. Accordingly, the investigators will access cortical excitability modulation measures in both depressed patients and healthy volunteers and compare their results. The investigators will also re-assess these measures after 6 weeks of antidepressant treatment. Finally, the investigators will study the association between cortical excitability measures and cognitive processes using an innovative cognitive task.

DETAILED DESCRIPTION:
Study objectives

The aim of this study is to evaluate differences in the modulation of cortical excitability by a repetitive Transcranial Magnetic Stimulation (rTMS) protocol between patients with Major Depressive Disorder (MDD) and healthy people. The investigators hypothesize that patients with MDD exhibit less modulation of cortical excitability when compared to healthy people.

In order to accomplish this goal the investigators will:

* Compare measures of cortical excitability between patients with MDD and healthy individuals;
* Compare the degree of modulation of cortical excitability in motor cortex after the application of rTMS, between healthy individuals and patients with MDD;
* Study the progression/evolution of these measures in the group of patients with MDD after 6 weeks of antidepressant treatment, while comparing patients that respond to treatment with patients with symptoms resistant to treatment;
* Analyze the relationship between cortical excitability measures and cortical excitability modulation. Study participants will perform a psychophysical task, on a computer game, in order to evaluate certain cognitive processes and understand if there are differences in performance between patients with depression and healthy subjects.

Data Collection

* Clinical assessment: Clinical interview will be performed with help of psychiatric, psychological and cognitive psychometric instruments (self-report questionnaires and structured interviews) to assess the participants' health.
* Behavioural assessment: Participants will perform a psychophysical task in the form of a computer game.
* Neurophysiological evaluation: protocol for assessing excitability and excitability modulation of the motor cortex by EMT and EMTr (ETBi).

Procedures

The participants recruited for the present project will be patients who are already being treated by health professionals at the Champalimaud Clinical Center, as well as healthy individuals, recruited from the nearby community. One cohort will include patients with active/symptomatic MDD and a second cohort will include patients with MDD in remission that are still in treatment. The third cohort will include a control group of healthy individuals. After they are referred to participate in this study, and if consent to participate is collected, they will be assessed to confirm their eligibility and group allocation will be performed. The study participants from all three observational groups will be submitted to (1) full clinical information assessment, (2) will be asked to perform a psychophysical task, i.e. a computer game. Finally, (3) the neurophysiological evaluation protocol will be applied. This neurophysiological evaluation protocol will be performed in two visits separated by at least 48h. This will make it possible to assess cortical excitability measures in both hemispheres independently and safely, allowing the acquisition of interhemispheric asymmetry measures. The order in which the cerebral hemispheres will be assessed will be randomized between participants. The first visit should take no longer than 120 minutes, and the second will last less than 45 minutes. Participants in the study will also be asked to come for a second study visit, to the Champalimaud Clinical Center, approximately 6 weeks after the first visit, the same study protocol will be repeated, in two consecutive sessions with the same procedures.Participants will not be rewarded monetarily; they will be supported for travel to the Clinical Center that may be necessary outside their individual clinical follow-up

ELIGIBILITY:
Inclusion criteria (clinical groups):

1. Diagnosis of major depressive episode or disorder as provided in the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) (American Psychiatric Association. 2013).

Exclusion criteria (clinical groups):

1. Moderate to severe suicide risk;
2. Known personal history of bipolar disorder or psychotic disorder;
3. Alcohol or other substance abuse and/or dependence;
4. Developmental disorder;
5. Dementia;
6. Presence of uncontrolled active medical illness;
7. Known structural lesion of the central nervous system;
8. Electrical or metallic brain implants;
9. Cardiac implants;
10. Epilepsy;
11. Active use of medication known to cause seizures;
12. Pregnancy;
13. Breastfeeding.

For the healthy control group, participants will also be recruited at the Champalimaud Clinical Center, by advertisement in places of public circulation. The recruitment of this population will be done in order to generate a pairing with both clinical groups in terms of age and sex. The same exclusion criteria will be applied, as well as the presence of any history of neuropsychiatric disease. The total number of participants for this study will be approximately 90 volunteers. Exclusion criteria will be assessed through self-report and/or MINI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be adults, aged 18 to 65 years, that will be recruited either for the clinical groups or healthy subjects group. The clinical population will include individuals with MDE diagnosis, and will be divided into two clinical groups:
  1. Patients in the acute phase of MDE, at the time they start a new antidepressant treatment (n≈30);
  2. Patients with symptomatic improvement, on continuation or maintenance antidepressant treatment (n≈30).
  All groups, including healthy subjects, will be paired by age and sex.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-05-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline left cortical excitability modulation | Baseline
  Differences between groups in left cortical excitability modulation at baseline. Left cortical excitability modulation will be computed by assessing motor evoked potentials (MEP) before and after left-sided TMS modulation protocol.

SECONDARY OUTCOMES:
Left cortical excitability modulation changes according to treatment response | Baseline and after ~6 weeks.
  Differences between responders and non responders to a new antidepressant treatment of left cortical excitability modulation changes between baseline and after 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Albino J Oliveira-Maia, MD, MPH, PhD, Principal Investigator — Champalimaud Foundation
Locations (1):
- Champalimaud Foundation, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Benussi A, Di Lorenzo F, Dell'Era V, Cosseddu M, Alberici A, Caratozzolo S, Cotelli MS, Micheli A, Rozzini L, Depari A, Flammini A, Ponzo V, Martorana A, Caltagirone C, Padovani A, Koch G, Borroni B. Transcranial magnetic stimulation distinguishes Alzheimer disease from frontotemporal dementia. Neurology. 2017 Aug 15;89(7):665-672. doi: 10.1212/WNL.0000000000004232. Epub 2017 Jul 26. PMID 28747446
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Chang WH, Fried PJ, Saxena S, Jannati A, Gomes-Osman J, Kim YH, Pascual-Leone A. Optimal number of pulses as outcome measures of neuronavigated transcranial magnetic stimulation. Clin Neurophysiol. 2016 Aug;127(8):2892-2897. doi: 10.1016/j.clinph.2016.04.001. Epub 2016 Apr 12. PMID 27156431
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Cincotta M, Giovannelli F, Borgheresi A, Balestrieri F, Toscani L, Zaccara G, Carducci F, Viggiano MP, Rossi S. Optically tracked neuronavigation increases the stability of hand-held focal coil positioning: evidence from "transcranial" magnetic stimulation-induced electrical field measurements. Brain Stimul. 2010 Apr;3(2):119-23. doi: 10.1016/j.brs.2010.01.001. Epub 2010 Jan 29. PMID 20633439
- [Background] Concerto C, Lanza G, Cantone M, Pennisi M, Giordano D, Spampinato C, Ricceri R, Pennisi G, Aguglia E, Bella R. Different patterns of cortical excitability in major depression and vascular depression: a transcranial magnetic stimulation study. BMC Psychiatry. 2013 Nov 9;13:300. doi: 10.1186/1471-244X-13-300. PMID 24206945
- [Background] Daskalakis ZJ, Farzan F, Barr MS, Maller JJ, Chen R, Fitzgerald PB. Long-interval cortical inhibition from the dorsolateral prefrontal cortex: a TMS-EEG study. Neuropsychopharmacology. 2008 Nov;33(12):2860-9. doi: 10.1038/npp.2008.22. Epub 2008 Mar 5. PMID 18322469
- [Background] Fitzgerald, Paul B., and Z. Jeff Daskalakis. Repetitive Transcranial Magnetic Stimulation Treatment for Depressive Disorders: A Practical Guide. Heidelberg: Springer, 2013.
- [Background] Fried PJ, Jannati A, Davila-Perez P, Pascual-Leone A. Reproducibility of Single-Pulse, Paired-Pulse, and Intermittent Theta-Burst TMS Measures in Healthy Aging, Type-2 Diabetes, and Alzheimer's Disease. Front Aging Neurosci. 2017 Aug 21;9:263. doi: 10.3389/fnagi.2017.00263. eCollection 2017. PMID 28871222
- [Background] Goldsworthy MR, Hordacre B, Ridding MC. Minimum number of trials required for within- and between-session reliability of TMS measures of corticospinal excitability. Neuroscience. 2016 Apr 21;320:205-9. doi: 10.1016/j.neuroscience.2016.02.012. Epub 2016 Feb 9. PMID 26872998
- [Background] Huang YZ, Rothwell JC. The effect of short-duration bursts of high-frequency, low-intensity transcranial magnetic stimulation on the human motor cortex. Clin Neurophysiol. 2004 May;115(5):1069-75. doi: 10.1016/j.clinph.2003.12.026. PMID 15066532
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Jahanshahi M, Ridding MC, Limousin P, Profice P, Fogel W, Dressler D, Fuller R, Brown RG, Brown P, Rothwell JC. Rapid rate transcranial magnetic stimulation--a safety study. Electroencephalogr Clin Neurophysiol. 1997 Dec;105(6):422-9. doi: 10.1016/s0924-980x(97)00057-x. PMID 9448643
- [Background] Julkunen P, Saisanen L, Danner N, Niskanen E, Hukkanen T, Mervaala E, Kononen M. Comparison of navigated and non-navigated transcranial magnetic stimulation for motor cortex mapping, motor threshold and motor evoked potentials. Neuroimage. 2009 Feb 1;44(3):790-5. doi: 10.1016/j.neuroimage.2008.09.040. Epub 2008 Oct 11. PMID 18976714
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Kim DR, Epperson N, Pare E, Gonzalez JM, Parry S, Thase ME, Cristancho P, Sammel MD, O'Reardon JP. An open label pilot study of transcranial magnetic stimulation for pregnant women with major depressive disorder. J Womens Health (Larchmt). 2011 Feb;20(2):255-61. doi: 10.1089/jwh.2010.2353. PMID 21314450
- [Background] Kupfer DJ, Frank E, Phillips ML. Major depressive disorder: new clinical, neurobiological, and treatment perspectives. Lancet. 2012 Mar 17;379(9820):1045-55. doi: 10.1016/S0140-6736(11)60602-8. Epub 2011 Dec 19. PMID 22189047
- [Background] Leykin Y, Roberts CS, Derubeis RJ. Decision-Making and Depressive Symptomatology. Cognit Ther Res. 2011 Aug;35(4):333-341. doi: 10.1007/s10608-010-9308-0. Epub 2010 May 4. PMID 21841849
- [Background] Loo CK, McFarquhar TF, Mitchell PB. A review of the safety of repetitive transcranial magnetic stimulation as a clinical treatment for depression. Int J Neuropsychopharmacol. 2008 Feb;11(1):131-47. doi: 10.1017/S1461145707007717. Epub 2007 Sep 20. PMID 17880752
- [Background] Machii K, Cohen D, Ramos-Estebanez C, Pascual-Leone A. Safety of rTMS to non-motor cortical areas in healthy participants and patients. Clin Neurophysiol. 2006 Feb;117(2):455-71. doi: 10.1016/j.clinph.2005.10.014. Epub 2006 Jan 4. PMID 16387549
- [Background] Maeda F, Keenan JP, Pascual-Leone A. Interhemispheric asymmetry of motor cortical excitability in major depression as measured by transcranial magnetic stimulation. Br J Psychiatry. 2000 Aug;177:169-73. doi: 10.1192/bjp.177.2.169. PMID 11026958
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Background] Oliveira-Maia AJ, Press D, Pascual-Leone A. Modulation of motor cortex excitability predicts antidepressant response to prefrontal cortex repetitive transcranial magnetic stimulation. Brain Stimul. 2017 Jul-Aug;10(4):787-794. doi: 10.1016/j.brs.2017.03.013. Epub 2017 Mar 31. PMID 28438543
- [Background] Player MJ, Taylor JL, Weickert CS, Alonzo A, Sachdev P, Martin D, Mitchell PB, Loo CK. Neuroplasticity in depressed individuals compared with healthy controls. Neuropsychopharmacology. 2013 Oct;38(11):2101-8. doi: 10.1038/npp.2013.126. Epub 2013 May 16. PMID 23676792
- [Background] Radhu, Natasha, Daniel M. Blumberger, and Zafiris J. Daskalakis. "Cortical Inhibition and Excitation in Neuropsychiatric Disorders Using Transcranial Magnetic Stimulation." In Transcranial Direct Current Stimulation in Neuropsychiatric Disorders, edited by André Brunoni, Michael Nitsche, and Colleen Loo, 85-102. Cham: Springer International Publishing, 2016. https://doi.org/10.1007/978-3-319-33967-2_6.
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Schrader LM, Stern JM, Koski L, Nuwer MR, Engel J Jr. Seizure incidence during single- and paired-pulse transcranial magnetic stimulation (TMS) in individuals with epilepsy. Clin Neurophysiol. 2004 Dec;115(12):2728-37. doi: 10.1016/j.clinph.2004.06.018. PMID 15546781
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Siebner HR, Hartwigsen G, Kassuba T, Rothwell JC. How does transcranial magnetic stimulation modify neuronal activity in the brain? Implications for studies of cognition. Cortex. 2009 Oct;45(9):1035-42. doi: 10.1016/j.cortex.2009.02.007. Epub 2009 Mar 3. PMID 19371866
- [Background] Vignaud P, Damasceno C, Poulet E, Brunelin J. Impaired Modulation of Corticospinal Excitability in Drug-Free Patients With Major Depressive Disorder: A Theta-Burst Stimulation Study. Front Hum Neurosci. 2019 Feb 26;13:72. doi: 10.3389/fnhum.2019.00072. eCollection 2019. PMID 30863297
- [Background] Wainwright SR, Galea LA. The neural plasticity theory of depression: assessing the roles of adult neurogenesis and PSA-NCAM within the hippocampus. Neural Plast. 2013;2013:805497. doi: 10.1155/2013/805497. Epub 2013 Apr 9. PMID 23691371
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057